CLINICAL TRIAL: NCT04998396
Title: A Phase 1/2 Open-Label Study of the Safety and Clinical Activity of Gene Therapy for Canavan Disease Through Administration of an Adeno-Associated Virus (AAV) Serotype 9-Based Recombinant Vector Encoding the Human ASPA Gene
Brief Title: A Study of AAV9 Gene Therapy in Participants With Canavan Disease (CANaspire Clinical Trial)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aspa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CVN-102
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Canavan Disease
Keywords: Canavan Disease; AAV; AAV9; Gene therapy; Aspartoacylase; ASPA; ASPA gene; rAAV9; ACY2; Aminoacylase 2; Spongy degeneration; N-acetyl-L-aspartic acid (NAA); N-acetylaspartate; Rare disease; Inherited Metabolic Disorders; Leukodystrophy; Leukoencephalopathies; Autosomal Recessive Disorder; Neurodevelopmental diseases; CANaspire Clinical Trial
MeSH Terms: conditions — Canavan Disease; Rare Diseases; Leukoencephalopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose-Finding Phase: BBP-812 Dose Level 1 (Cohort 1) (Experimental): Participants will receive a single intravenous (IV) infusion of low-dose BBP-812 on Day 0 in the dose-finding phase of the study.
  Interventions: Biological: AAV9 BBP-812
- Dose-Finding Phase: BBP-812 Dose Level 2 (Cohort 2) (Experimental): Participants will receive a single IV infusion of high-dose BBP-812 on Day 0 in the dose-finding phase of the study.
  Interventions: Biological: AAV9 BBP-812
- Enrollment Expansion Phase: BBP-812 (Experimental): Participants will receive a single IV infusion of BBP-812 at the selected dose from the dose-finding phase on Day 0 in expansion phase of the study.
  Interventions: Biological: AAV9 BBP-812

INTERVENTIONS:
Biological: AAV9 BBP-812 — Sterile solution for injection for 1-time use via volumetric infusion pump

SUMMARY:
The main objective of this trial is to evaluate the safety, tolerability, and pharmacodynamic activity of BBP-812, an investigational AAV9-based gene therapy, in pediatric participants with Canavan disease.

DETAILED DESCRIPTION:
Canavan disease is an ultra-rare, profoundly disabling and fatal disease with no approved therapy. The Sponsor is developing BBP-812, an investigational gene therapy product for systemic delivery in participants with Canavan disease. BBP-812 is a recombinant adeno-associated virus serotype 9 (rAAV9) vector engineered to deliver the aspartoacylase (ASPA) transgene under control of a ubiquitous promoter to restore ASPA expression in both neuronal and non-neuronal cell types.

ELIGIBILITY:
Key Inclusion Criteria:

* Maximum age for inclusion is 30 months.
* Participant has stable health in the opinion of the investigator and as confirmed by medical history and laboratory studies with no acute or chronic hematologic, renal, liver, immunologic, or neurologic disease (other than Canavan disease).
* Participant has biochemical, genetic, and clinical diagnosis of Canavan disease:

  * Elevated urinary NAA and
  * Biallelic mutation of the ASPA gene determined at Screening or documented in the participant's medical history.
  * Active clinical signs of Canavan disease
* Participant is up to date on all immunizations per local guidelines

Key Exclusion Criteria:

* Tests positive for total anti-AAV9 antibodies determined by enzyme-linked immunosorbent assay (ELISA).
* Received prior gene therapy or other therapy (including vaccines) involving AAV.
* Participant is receiving high-dose therapy with immunosuppressants.
* Participant has significantly progressed Canavan disease characterized as:

  * Presence of continuous/constant decerebrate or decorticate posturing,
  * Recurrent status epilepticus, or
  * Recalcitrant seizures that do not respond while on 3 or more anti-epileptic medications

Max Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2030-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline up to Week 52
Change from Baseline to 12 Months Post-Infusion in Urine N-acetylaspartate (NAA) Levels | Baseline, Month 12
Change from Baseline to 12 Months Post-Infusion in Central Nervous System (CNS) NAA, as Measured by Magnetic Resonance Spectroscopy (MRS) | Baseline, Month 12

SECONDARY OUTCOMES:
Change from Baseline to Week 52 in Gross Motor Assessment, Gross Motor Function Measure-88 | Baseline, Week 52
Change from Baseline to Week 52 in Fine Motor Assessment, Bayley-4 | Baseline, Week 52
Change from Baseline to Week 52 in Cognitive Assessment, Bayley-4 | Baseline, Week 52
Change from Baseline to Week 52 in Communication Assessment, Bayley-4 | Baseline, Week 52
Change from Baseline to Week 52 in Adaptive Function, Vineland-3 | Baseline, Week 52

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Massachusetts General Hospital (MGH); Center for Rare Neurological Diseases (CRND), Boston, Massachusetts
  - Weill Cornell Medicine; Division of Pediatric Neurology, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aspa Therapeutics Company Website — http://aspatx.com
- See also: CANaspire Clinical Trial Website — https://treatcanavan.com/canaspire-trial/